CLINICAL TRIAL: NCT03097679
Title: Self-expanding Nitinol Stents of High vs. Low Chronic Outward Force in De-novo Femoropopliteal Occlusive Arterial Lesions
Acronym: BIOFLEX-COF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alexander Wressnegger, Dr.med.univ., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1026/2015
Record Dates: First submitted 2017-03-14; First posted 2017-03-31 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Stent Restenosis; Intimal Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low COF-group (Active Comparator): The low COF-group receives a thin-strut stent (Pulsar, Biotronik AG, Bülach, Switzerland) with minimal oversizing (according to manufacturer's Instructions For Use)
  Interventions: Device: Pulsar Stent
- high COF-group (Active Comparator): The high COF-group receives a stiffer-stent (Lifestent Flexstar, Bard Peripheral Vascular Inc., Tempe, AZ, USA) with maximal oversizing (according to manufacturer's Instructions For Use).
  Interventions: Device: LifeStent Flexstar Vascular Stent

INTERVENTIONS:
Device: Pulsar Stent — Percutane transluminal stent angioplasty with a Pulsar Stent of the superficial femoral artery for the treatment of peripheral arterial occlusive disease.
  Arms: low COF-group
Device: LifeStent Flexstar Vascular Stent — Percutane transluminal stent angioplasty with a LifeStent Flexstar Vascular Stent of the superficial femoral artery for the treatment of peripheral arterial occlusive disease.
  Arms: high COF-group

SUMMARY:
The objective of the BIOFLEX-COF trial is to investigate differences in formation of intimal hyperplasia at one and two years after implantation of nitinol-stents with high vs. low COF in de-novo femoropopliteal occlusive lesions in patients with symptomatic peripheral arterial disease.

The BIOFLEX-COF trial is a prospective, randomized controlled trial. 80 subjects will be enrolled and randomly assigned to either a high COF group (LifeStent Vascular Stent) or low COF group (Pulsar).

DETAILED DESCRIPTION:
Self-expanding nitinol stents must be oversized at least by a minimal amount to ensure contact with the vessel wall and prevent migration. Once the stent is deployed it exerts a continuous force upon the vascular wall, termed chronic outward force (COF). Data about COF and neointimal hyperplasia in humans are currently lacking. Some animal studies, though, found a markedly increased neointimal hyperplasia in stents with high oversizing and thus high COF. The objective of the BIOFLEX-COF trial is to investigate differences in formation of intimal hyperplasia at one and two years after implantation of nitinol-stents with high vs. low COF in de-novo femoropopliteal occlusive lesions in patients with symptomatic peripheral arterial disease.

The BIOFLEX-COF trial is a prospective, randomized controlled trial. 80 subjects will be enrolled and randomly assigned to either a high COF group (LifeStent Vascular Stent) or low COF group (Pulsar). Diameter of implanted stents will be measured at every two millimetres along the stent axis on DICOM images of the respective completion angiography using image processing software.

The scheduled time for recruitment is 2 years. There will be two follow-up evaluations at 12 and 24 months.

Primary endpoint is the amount of in-stent neointima at one year, assessed by contrast-enhanced CT angiography (CTA). Secondary objectives are the amount of in-stent neointima at two years, device- and procedure-related adverse events and target lesion revascularisation (TLR) rate.

In the control examinations stent diameter and true lumen diameter will be measured on DICOM images every two millimetres along the stent axis to quantify the relative amount of in-stent restenosis.

The present study is challenging in that it compares two different self-expanding nitinol-stents head-to-head against each other. To optimize the power of this study, both clinical TLR and binary re-stenosis at Colour flow Doppler Ultrasound were dropped as primary endpoints. Instead the amount of neointima inside the stent accessed by CTA was selected as outcome parameter.

The study differs further from similar previous trials in its generous inclusions criteria. This was done in effort to perform the trial on a patient sample that closely represents real-world patients of a specialised endovascular centre.

ELIGIBILITY:
Inclusion Criteria:

Patient related:

1. Subject (or their legal guardian) has read, understood and provided written informed consent, which has been reviewed and approved by the Institutional Review Board.
2. At least 18 years of age.
3. Male, infertile female or female participants of child bearing potential practicing an acceptable method of birth control with a negative pregnancy test within 7-days prior to study procedure.
4. Projected life expectancy of greater than two years.
5. The ability to comply with protocol follow-up requirements and required testing.

Clinical:

1. Lifestyle-limiting claudication or CLI (meeting angiographic entry criteria) affecting a lower extremity (Rutherford stages 2-5). Patients with Rutherford stage 2 are only eligible after unsuccessful conventional and/or medicamentous therapy.
2. Resting ankle-brachial index (ABI) ≤ 0.8 in the study limb.
3. Inflow lesion - if present - has been treated successfully (inflow treatment in same procedure permissible)

Angiographic and Lesion Requirements (assessed intraoperatively):

1. TASC A-D lesions from stenoses /occlusions ≤ 35cm.
2. Popliteal artery is patent 5 cm proximal to the radiographic knee joint line.
3. Reference diameter of 4.0 - 7.0 mm in proximal and distal treatment segments within the SFA.
4. Patent SFA orifice (the proximal 5 mm after femoral bifurcation).
5. At least one patent (<50% stenotic) inflow vessel present, proven angiographically. Study eligibility is given when inflow lesion has been treated successfully (inflow treatment in same procedure permissible). Successful treatment of inflow lesion is defined as <50% stenosis without death or severe vascular complication.
6. At least one patent (<50% stenotic)tibial artery runoff to the ankle present, proven angiographically. Study eligibility is given when runoff vessel lesion has been treated successfully (inflow treatment in same procedure permissible). Successful treatment of inflow lesion is defined as <50% stenosis without death or severe vascular complication.Guidewire has successfully traversed lesion and is within the true lumen of the distal vessel.

Exclusion Criteria:

1. Pregnant and/or breast-feeding women.
2. Lesion length > 35 cm.
3. Flow-limiting occlusive disease of inflow and / or outflow arteries that cannot be treated sufficiently.
4. Previous stenting or femoral bypass surgery in the target vessel.
5. Clinical relevant aneurysmatic disease of the abdominal aorta, ipsilateral femoral arteries or arteries of the knee.
6. Rutherford stage 0, 1 or 6
7. Non-atherosclerotic disease resulting in occlusion (e.g., embolism, Buerger's disease, vasculitis).
8. Septicaemia.
9. Ischemic stroke within the last three months.
10. Any previously known coagulation disorder, including hypercoagulability
11. Morbid obesity or operative scarring that precludes percutaneous approach (physician's discretion).
12. Contraindication to anticoagulation or antiplatelet therapy.
13. Known allergy to medication or contrast media used in this trial, if pre-treatment is not possible (physician's discretion).
14. Known allergies to stent components (especially Nickel).
15. Severe calcification of the target lesion.
16. Current participation in another clinical research trial, that has not reached its primary endpoint.
17. The patient is institutionalized based on a legal verdict.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Amount of in-stent restenosis | one and two years post-procedure
  Mean amount of in-stent restenosis in percent along the stent axis at one and two years post-procedure.

SECONDARY OUTCOMES:
Adverse Events ISO 14155:2011 | within two years post-procedure
  Adverse Events ISO 14155:2011
Target lesion revascularisation (TLR) | within two years post-procedure
  In patients with TLR the amount of in-stent restenosis will be assessed at the time of TLR.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lammer J, Zeller T, Hausegger KA, Schaefer PJ, Gschwendtner M, Mueller-Huelsbeck S, Rand T, Funovics M, Wolf F, Rastan A, Gschwandtner M, Puchner S, Beschorner U, Ristl R, Schoder M. Sustained benefit at 2 years for covered stents versus bare-metal stents in long SFA lesions: the VIASTAR trial. Cardiovasc Intervent Radiol. 2015 Feb;38(1):25-32. doi: 10.1007/s00270-014-1024-9. Epub 2014 Dec 5. PMID 25472936
- [Background] Jaff MR, White CJ, Hiatt WR, Fowkes GR, Dormandy J, Razavi M, Reekers J, Norgren L. An Update on Methods for Revascularization and Expansion of the TASC Lesion Classification to Include Below-the-Knee Arteries: A Supplement to the Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II): The TASC Steering Comittee(.). Ann Vasc Dis. 2015;8(4):343-57. doi: 10.3400/avd.tasc.15-01000. Epub 2015 Oct 23. PMID 26730266
- [Background] Saxon RR, Dake MD, Volgelzang RL, Katzen BT, Becker GJ. Randomized, multicenter study comparing expanded polytetrafluoroethylene-covered endoprosthesis placement with percutaneous transluminal angioplasty in the treatment of superficial femoral artery occlusive disease. J Vasc Interv Radiol. 2008 Jun;19(6):823-32. doi: 10.1016/j.jvir.2008.02.008. Epub 2008 Apr 10. PMID 18503895
- [Background] Rastan A, Krankenberg H, Baumgartner I, Blessing E, Muller-Hulsbeck S, Pilger E, Scheinert D, Lammer J, Beschorner U, Noory E, Neumann FJ, Zeller T. Stent placement vs. balloon angioplasty for popliteal artery treatment: two-year results of a prospective, multicenter, randomized trial. J Endovasc Ther. 2015 Feb;22(1):22-7. doi: 10.1177/1526602814564386. PMID 25775675
- [Background] Dick P, Wallner H, Sabeti S, Loewe C, Mlekusch W, Lammer J, Koppensteiner R, Minar E, Schillinger M. Balloon angioplasty versus stenting with nitinol stents in intermediate length superficial femoral artery lesions. Catheter Cardiovasc Interv. 2009 Dec 1;74(7):1090-5. doi: 10.1002/ccd.22128. PMID 19859954
- [Background] Krankenberg H, Schluter M, Steinkamp HJ, Burgelin K, Scheinert D, Schulte KL, Minar E, Peeters P, Bosiers M, Tepe G, Reimers B, Mahler F, Tubler T, Zeller T. Nitinol stent implantation versus percutaneous transluminal angioplasty in superficial femoral artery lesions up to 10 cm in length: the femoral artery stenting trial (FAST). Circulation. 2007 Jul 17;116(3):285-92. doi: 10.1161/CIRCULATIONAHA.107.689141. Epub 2007 Jun 25. PMID 17592075
- [Background] Dake MD, Ansel GM, Jaff MR, Ohki T, Saxon RR, Smouse HB, Zeller T, Roubin GS, Burket MW, Khatib Y, Snyder SA, Ragheb AO, White JK, Machan LS; Zilver PTX Investigators. Paclitaxel-eluting stents show superiority to balloon angioplasty and bare metal stents in femoropopliteal disease: twelve-month Zilver PTX randomized study results. Circ Cardiovasc Interv. 2011 Oct 1;4(5):495-504. doi: 10.1161/CIRCINTERVENTIONS.111.962324. Epub 2011 Sep 27. PMID 21953370
- [Background] Deloose K, Lauwers K, Callaert J, Maene L, Keirse K, Verbist J, Peeters P, Bosiers M. Drug-eluting technologies in femoral artery lesions. J Cardiovasc Surg (Torino). 2013 Apr;54(2):217-24. PMID 23558657
- [Background] Brodmann M. Prime time for drug eluting balloons in SFA interventions? J Cardiovasc Surg (Torino). 2014 Aug;55(4):461-4. Epub 2014 Jun 18. PMID 24941235
- [Background] Minar E, Schillinger M. Innovative technologies for SFA occlusions: drug coated balloons in SFA lesions. J Cardiovasc Surg (Torino). 2012 Aug;53(4):481-6. PMID 22854528
- [Background] Schmidt W, Wissgott C, Andresen R, Behrens P, Schmitz KP. Performance characteristics of modern self-expanding nitinol stents indicated for SFA. Rofo. 2011 Sep;183(9):818-25. doi: 10.1055/s-0031-1273445. Epub 2011 Jul 12. PMID 21751121
- [Background] Johnston CR, Lee K, Flewitt J, Moore R, Dobson GM, Thornton GM. The mechanical properties of endovascular stents: an in vitro assessment. Cardiovasc Eng. 2010 Sep;10(3):128-35. doi: 10.1007/s10558-010-9097-9. PMID 20717726
- [Background] Cho H, Nango M, Sakai Y, Sohgawa E, Kageyama K, Hamamoto S, Kitayama T, Yamamoto A, Miki Y. Neointimal hyperplasia after stent placement across size-discrepant vessels in an animal study. Jpn J Radiol. 2014 Jun;32(6):340-6. doi: 10.1007/s11604-014-0311-3. Epub 2014 Apr 9. PMID 24715330
- [Background] Zhao HQ, Nikanorov A, Virmani R, Jones R, Pacheco E, Schwartz LB. Late stent expansion and neointimal proliferation of oversized Nitinol stents in peripheral arteries. Cardiovasc Intervent Radiol. 2009 Jul;32(4):720-6. doi: 10.1007/s00270-009-9601-z. Epub 2009 May 30. PMID 19484292
- [Background] Freeman JW, Snowhill PB, Nosher JL. A link between stent radial forces and vascular wall remodeling: the discovery of an optimal stent radial force for minimal vessel restenosis. Connect Tissue Res. 2010 Aug;51(4):314-26. doi: 10.3109/03008200903329771. PMID 20388019
- [Background] Saguner AM, Traupe T, Raber L, Hess N, Banz Y, Saguner AR, Diehm N, Hess OM. Oversizing and restenosis with self-expanding stents in iliofemoral arteries. Cardiovasc Intervent Radiol. 2012 Aug;35(4):906-13. doi: 10.1007/s00270-011-0275-y. Epub 2011 Oct 18. PMID 22006026
- [Background] Kirsch EC, Khangure MS, Morling P, York TJ, McAuliffe W. Oversizing of self-expanding stents: influence on the development of neointimal hyperplasia of the carotid artery in a canine model. AJNR Am J Neuroradiol. 2002 Jan;23(1):121-7. PMID 11827884
- [Background] Vorwerk D, Redha F, Neuerburg J, Clerc C, Gunther RW. Neointima formation following arterial placement of self-expanding stents of different radial force: experimental results. Cardiovasc Intervent Radiol. 1994 Jan-Feb;17(1):27-32. doi: 10.1007/BF00197911. PMID 8187129
- [Background] Saxon RR, Chervu A, Jones PA, Bajwa TK, Gable DR, Soukas PA, Begg RJ, Adams JG, Ansel GM, Schneider DB, Eichler CM, Rush MJ. Heparin-bonded, expanded polytetrafluoroethylene-lined stent graft in the treatment of femoropopliteal artery disease: 1-year results of the VIPER (Viabahn Endoprosthesis with Heparin Bioactive Surface in the Treatment of Superficial Femoral Artery Obstructive Disease) trial. J Vasc Interv Radiol. 2013 Feb;24(2):165-73; quiz 174. doi: 10.1016/j.jvir.2012.10.004. Epub 2013 Jan 28. PMID 23369553
- [Background] Goueffic Y, Kaladji A, Guyomarch B, Montagne C, Fairier D, Gestin S, Riche VP, Vent PA, Chaillou P, Costargent A, Patra P. Bare metal stent versus paclitaxel eluting stent for intermediate length femoropopliteal arterial lesions (BATTLE trial): study protocol for a randomized controlled trial. Trials. 2014 Oct 30;15:423. doi: 10.1186/1745-6215-15-423. PMID 25359394
- [Derived] Wressnegger A, Kaider A, Funovics MA. Self-expanding nitinol stents of high versus low chronic outward force in de novo femoropopliteal occlusive arterial lesions (BIOFLEX-COF trial): study protocol for a randomized controlled trial. Trials. 2017 Dec 14;18(1):594. doi: 10.1186/s13063-017-2338-0. PMID 29237489